CLINICAL TRIAL: NCT03522142
Title: A Phase 1a/1b Study Exploring the Safety and Tolerability of INCB081776 in Participants With Advanced Malignancies
Brief Title: A Study Exploring the Safety and Tolerability of INCB081776 in Participants With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated after careful review of the overall clinical activity of this compound and a lack of robust efficacy. The study closure is not based on safety concerns.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 81776-101; 2023-504499-29-00 (Registry Identifier: EU CT Number); 2020-004867-26 (EudraCT Number)
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors; AXL; MER; AXL/MER; PD-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INCB081776 (Experimental): Single-agent INCB081776.
  Interventions: Drug: INCB081776
- INCB081776 + INCMGA00012 (Experimental): INCB081776 in combination with INCMGA00012.
  Interventions: Drug: INCB081776; Drug: INCMGA00012

INTERVENTIONS:
Drug: INCB081776 — INCB081776 administered once or twice daily orally with water after a fast of at least 2 hours before and at least 1 hour after the dose.
Drug: INCMGA00012 — INCMGA0012 administered intravenously according to the label as 500 mg every 4 weeks
  Other Names: retifanlimab
  Arms: INCB081776 + INCMGA00012

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, pharmacokinetics, pharmacodynamics, and early clinical activity of single-agent INCB081776 (Part 1) and INCB081776 in combination with INCMGA00012 (Part 2).

ELIGIBILITY:
Inclusion Criteria:

• Male and female participants at least 18 years of age with advanced malignancies who have received or been intolerant to standard therapy:

Parts 1A and 2A:

* Histologically confirmed advanced or metastatic gastric or GEJ adenocarcinoma, HCC, melanoma, NSCLC, RCC, soft-tissue sarcoma, SCCHN (recurrent or metastatic), TNBC, or urothelial carcinoma. Additional tumor histologies, including MSI-H tumors, may be allowed with approval from the medical monitor.
* Measurable disease per RECIST v1.1.

Parts 1B and 2B:

• Histologic confirmation of the cohort-specific tumor types specified below: Cohort 1 - Advanced or metastatic melanoma Cohort 2 - Advanced or metastatic NSCLC Cohort 3 - Recurrent or metastatic SCCHN Cohort 4 - Advanced or metastatic soft-tissue sarcoma

* Cohorts 1-3 must have received 1 prior PD-1/L1 treatment and have experienced PD during or after that treatment and have progressed on other SOC therapy(ies); Cohort 4 must be PD-1/L1 treatment naïve but have progressed on SOC therapy(ies).
* Measurable disease per RECIST v1.1.
* Must be willing to submit to a fresh baseline tumor biopsy and an on-treatment biopsy between Cycle 2 Day 1 and Cycle 3 Day 1.
* Care should be taken to biopsy the same lesion for the baseline and on-treatment samples. If a participant has a solitary target lesion, this should not be biopsied.

Part 1C:

* Participants with relapsed/refractory AML following standard therapy; acute promyelocytic leukemia (M3) and therapy-related AML are excluded.
* FLT3-ITD and IDH1/2 wild-type or mutated are eligible; appropriate targeted therapy for participants with actionable mutations must have been received.

Exclusion Criteria:

* Laboratory values not within the protocol-defined range.
* History of retinal disease as defined in the protocol.
* Clinically significant cardiac disease as per protocol-defined criteria.
* History or presence of an ECG that, in the investigator's opinion, is clinically meaningful as per protocol-defined criteria.
* Untreated brain or central nervous system (CNS) metastases or brain or CNS metastases that have progressed as per protocol-defined criteria.
* Active or inactive autoimmune disease or syndrome that has required systemic treatment in the past 2 years or receiving systemic therapy for an autoimmune or inflammatory disease.
* Prior Grade 3 or higher immune-related AEs or any ocular toxicity on prior immunotherapy as per protocol-defined criteria.
* Receipt of any vitamin K antagonists, systemic corticosteroids, live vaccines, or treatment with any anticancer medications or investigational drugs within the protocol-defined intervals.
* Has not recovered to ≤ Grade 1 or baseline from toxic effects of prior therapy and/or complications from prior surgical intervention before starting study treatment.
* Active infection requiring systemic therapy.
* Evidence of hepatitis B virus or hepatitis C virus infection or risk of reactivation.
* Known history of HIV (HIV 1/2 antibodies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Part 1 (1A and 1B): Number of treatment-emergent adverse events (TEAEs) | Screening through 90 days after end of treatment, up to approximately 1 year.
  A TEAE is any adverse event (AE) either reported for the first time or worsening of a pre-existing event after first dose of study drug.
Part 1 (1A and 1B): Recommended Dose for Expansion (RDE) | Up to one year
  Recommended dose as a monotherapy as measured by safety, PK and data
Part 2 (2A & 2B): Number of treatment-emergent adverse events | Screening through 90 days after end of treatment, up to approximately 1 year
  A TEAE is any adverse event (AE) either reported for the first time or worsening of a pre-existing event after first dose of study drug.
Part 2 (2A & B): RDE in combination with INCMGA00012 | Up to one year
  Recommended dose as a combination as measured by safety, PK and data

SECONDARY OUTCOMES:
Part 1 and Part 2: Cmax of INCB081776 | Up to approximately 3 weeks.
  Maximum observed plasma concentration.
Part 1 and Part 2: Tmax of INCB081776 | Up to approximately 3 weeks.
  Time to maximum plasma concentration.
Part 1 and Part 2: t½ of INCB081776 | Up to approximately 3 weeks.
  Apparent plasma terminal phase disposition half-life
Part 1 and Part 2: Pharmacokinetic/ pharmacodynamic correlation | Up to approximately 3 weeks.
  To evaluate the correlation pharmacokinetic and pharmacodynamics of INCB081176
Part 1 and Part 2: Overall response rate | Up to approximately 1 year.
  Defined as the percentage of participants having complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Part 1 and Part 2: Disease control rate | Up to approximately 1 year.
  Defined as the percentage of participants having CR, PR, or stable disease (SD) per RECIST v1.1.
Part 1 and Part 2: Duration of response | Up to approximately 1 year.
  Defined as the time from earliest date of disease response until the earliest date of disease progression (per RECIST v1.1) or death due to any cause, if occurring sooner than progression.
Part 1 and Part 2: AUC0-t of INCB081776 | Up to approximately 3 weeks.
  Area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
Part 1 and Part 2: Cmin of INCB081776 | Up to approximately 3 weeks.
  Trough concentration of INCB081776
Part 1 and Part 2: AUC0-∞ of INCB081776 | Up to approximately 3 weeks.
  Area under the single-dose plasma concentration-time curve from Hour 0 to infinity
Part 1 and Part 2 : CL/F of INCB081776 | Up to approximately 3 weeks.
  Oral dose clearance
Part 1 and Part 2 : λz of INCB081776 | Up to approximately 3 weeks.
  Terminal elimination rate constant
Part 1 and Part 2 : Vz/F of INCB081776 | Up to approximately 3 weeks.
  Apparent oral dose volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Diane Hershock, MD, Study Director — Incyte Corporation
Locations (18):
- United States (9):
  - Yale Cancer Center, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Denmark (2):
  - Rigshospitalet Uni of Hospital of Copenhagen, Copenhagen
  - Odense University Hospital, Odense C
- Netherlands (3):
  - Netherlands Cancer Institute Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Utprøvingsenheten, Oslo University Hospital Radiumhospitalet, Oslo
- Sweden (2):
  - Skane University Hospital Lund, Lund
  - Karolinska University Hospital Solna, Stockholm

IPD SHARING:
Plan to Share IPD: No